CLINICAL TRIAL: NCT06165822
Title: A Phase I Study to Evaluate Drug-Drug Interaction of TQB3909 Tablets
Brief Title: A Study to Evaluate Drug-Drug Interaction of TQB3909 Tablets
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB3909-I-02
Record Dates: First submitted 2023-11-30; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Advanced Malignant Neoplasm
Keywords: Drug drug interaction
MeSH Terms: interventions — Itraconazole; Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Itraconazole drug-durg interaction (DDI) (Experimental): Itraconazole capsules, 0.2g once daily from Day 3 to Day 10 TQB3909 tablets, single oral dose on Day 1 and Day 8.
  Interventions: Drug: TQB3909 tablets; Drug: Itraconazole capsule
- Rifampicin DDI (Experimental): Rifampicin capsule, 0.6g once daily from Day 3 to Day 11. TQB3909 tablets, single oral dose on Day 1 and Day 10.
  Interventions: Drug: TQB3909 tablets; Drug: Rifampicin capsule

INTERVENTIONS:
Drug: TQB3909 tablets — TQB3909 100mg/tablet.
Drug: Itraconazole capsule — Itraconazole capsule is a strong inhibitor of CYP3A4.
  Arms: Itraconazole drug-durg interaction (DDI)
Drug: Rifampicin capsule — Rifampicin capsule is a strong inducer of CYP3A4.
  Arms: Rifampicin DDI

SUMMARY:
This is a single-center, open, single-dose, self-controlled phase I clinical trial to evaluate the effects of Itraconazole Capsules/Rifampicin Capsules on pharmacokinetics of TQB3909 tablets in vivo, and the safety of TQB3909 tablets and combined with Itraconazole Capsules/Rifampicin Capsules after single oral dose.

ELIGIBILITY:
Inclusion Criteria:

* At the time of signing the informed consent, males or females of between 18 and 45 years of age;
* Female weight ≥45 kg, male weight ≥50 kg, with a body mass index (BMI) between 19 and 26 kg/m2.
* Subjects in good health, as determined by a medical history, vital signs, physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory evaluations;
* Subjects can comply with the study procedures, voluntarily participate in the study, and sign the informed consent in person.

Exclusion Criteria:

* Subjects: pre-existing or existing circulatory system, endocrine system, nervous system, digestive system, respiratory system, genitourinary system, hematology, immunology, psychiatry and metabolic disorders mental diseases or abnormalities, or related chronic or acute diseases, which were not appropriate to participate in the trial as assessed by the investigators ;
* Subjects with systemic/local acute infection presented before study drug administration;
* Subjects who have a history of specific allergies, or allergies;
* Subjects who have difficulty in swallowing or have any gastrointestinal disorder that affects drug absorption at the time of screening；
* Subjects who cannot receive venous indwelling needle for blood sample collection；
* Subjects who cannot tolerate venous puncture or have a history of needle or blood sickness;
* Subjects who drank regularly within the 6 months prior to the first dosing, such as those who drank more than 14 units of alcohol per week or who had a positive alcohol breath test at the time of screening；
* Subjects who had a history of major surgery, had taken the study drug, or had participated in other drug clinical trials within 3 months prior to the first dosing；
* Subjects who donated blood or lost significant amounts of blood within 3 months prior to the first dosing；
* Subjects who had used drugs within 3 months prior to the first dosing, or tested positive for drugs, or had a history of drug abuse within 5 years prior to screening；
* Subjects who smoked more than 5 cigarettes per day within the 3 months prior to the first dosing or who could not stop using any tobacco products during the trial；
* Subjects who consumed excessive amounts of tea, coffee, and/or caffeinated beverages daily within the 30 days prior to the first dosing；
* Subjects who have used any drug that inhibits or induces liver metabolism of the drug within the 30 days prior to the first dosing；
* Subjects who have taken any prescription, over-the-counter, herbal, or health product within the 14 days prior to the first dosing；
* Subjects who have taken a special diet or other factors affecting drug absorption, distribution, metabolism, or excretion within 7 days prior to the first dosing；
* Subjects who ingested chocolate, any caffeinated, or xanthine-rich food or drink within 48 hours before the first dosing；
* Subjects who have special dietary requirements and cannot follow a uniform diet；
* Female subjects of child-bearing potential；
* Subjects judged by the investigators to be unsuitable to participate.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Inhibitor group: pre-dose, 1, 2, 3, 4, 5, 6, 7, 8, 10, 14, 24, 48, 72 hours (only on Day 8) after dose on Day 1 and Day 8. Inducer group: pre-dose, 1, 2, 3, 4, 5, 6, 7, 8, 10, 14, 24, 48 hours after dose on Day 1 and Day 10.
  Time to reach maximum (peak) plasma concentration following drug administration.
Maximum Plasma Concentration (Cmax) | Inhibitor group: pre-dose, 1, 2, 3, 4, 5, 6, 7, 8, 10, 14, 24, 48, 72 hours (only on Day 8) after dose on Day 1 and Day 8. Inducer group: pre-dose, 1, 2, 3, 4, 5, 6, 7, 8, 10, 14, 24, 48 hours after dose on Day 1 and Day 10.
  The maximum observed plasma concentration of TQB3909
Elimination half-life (t1/2) | Inhibitor group: pre-dose, 1, 2, 3, 4, 5, 6, 7, 8, 10, 14, 24, 48, 72 hours (only on Day 8) after dose on Day 1 and Day 8. Inducer group: pre-dose, 1, 2, 3, 4, 5, 6, 7, 8, 10, 14, 24, 48 hours after dose on Day 1 and Day 10.
  The time required for half of the drug to be eliminated from the plasma.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 12 days.
  Incidence of adverse events (AEs) based on the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- The First People's Hospital of Changzhou, Changzhou, Jiangsu, China